CLINICAL TRIAL: NCT05765539
Title: Performance of the Echopen Probe in Its Clinical Use for Pregnancy Follow-up in Senegal
Acronym: PRESTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: echOpen Factory (Industry)
Collaborators: Institut Pasteur de Dakar (Other); Fondation Sanofi Espoir (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-P01
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related
Keywords: Medical Device; Handheld Ultrasound; Echostethoscopy

STUDY DESIGN:
Intervention Model Description: A single group, comparative, non-randomized, controlled study. Each patient represents her/his own control: the patient is examined consecutively with the echOpen probe, then with the probe used in the department.
Masking Description: Midwife 'A' will begin by using either the echOpen probe or the classic US machine (in a random order, via sealed envelopes), and will then carry out the other type of examination. The results book will be filled in and validated after each examination, and it will not be possible to modify the results after the 2nd examination has been carried out. Another midwife (midwife 'B') will examine with the echOpen probe (blind to the first midwife's result). The alternation between midwife 'A' and midwife 'B' will also be random.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pregnant women benefitting ultrasound examination (Experimental): This is the unique arm of the study. This arm is made of eligible pregnant women, with a pregnancy of at least 37 weeks.
  Interventions: Device: echOpen O1 Handheld Ultrasound device

INTERVENTIONS:
Device: echOpen O1 Handheld Ultrasound device — The performance of the Handheld ultrasound device (echOpen O1 device) will be assessed during these visits for all evaluation criteria.
  * One examination with the US machine by the midwife focused on 4 targets ;
  * One examination with a classic US machine by the same midwife (comparator) including the search for the four targets ;
  * One examination with the US machine by a second operator ; Review of the images obtained by the US machine by the referring radiologist at a separate point of time.
  The mode of delivery and the vital status of the mother and newborn will also be collected.
  Operator A will start by using either the echOpen O1 device or the US machine (random order, via sealed envelopes) and will then perform the other type of examination.
  Another operator (Operator B) will come to perform an examination with the Handheld ultrasound device (blind to the result of the first operator).
  The switch between operators A and B will also be random.
  Other Names: Multicentric prospective comparative study

SUMMARY:
Pregnancy follow-up in a country with limited resources in decentralized areas usually consists of a clinical examination exclusively because of a lack of access to additional examination equipment and qualified personnel to use them. However, the pregnancy follow-up relies in part on the visual investigation by ultrasound scanners that estimate the risks of morbi-mortality for the mother and child during and after pregnancy. The WHO recommendations support at least one ultrasound before 24 weeks of amenorrhea. Thus, at the same time as a usual clinical examination, the possibility of visually assessing certain relevant criteria would help to increase the effectiveness of follow-up visits without complicating the care journey. A simple ultra-portable device would be an opportunity for caregivers to facilitate the detection of complications and thus offer a more adapted follow-up and orientation.

This would allow, in contexts where resources are limited, to improve monitoring and limit the risks of complications due to inappropriate management.

DETAILED DESCRIPTION:
The echOpen O1 Ultrasound Probe is a medical device designed to guide the diagnosis during clinical examination by providing a non-invasive, non-irradiant inside body image.

The investigator's hypothesis is that the use of this ultrasound stethoscopy probe during pregnancy, by a trained midwife, would improve the development and outcome of pregnancy for women by identifying situations requiring specificity. Through this protocol, the investigators propose a pilot study to evaluate, under field conditions, the performance of the echOpen O1 probe as part of the 3rd-trimester pregnancy monitoring, compared to a standard ultrasound examination, routinely performed with an ultrasound machine.

The main objective of this prospective pilot study is to evaluate the performance and operationality of the echOpen O1 probe from the 37th week of amenorrhea.

The secondary objectives are :

* To evaluate the feasibility and usability of the echOpen O1 probe in the context of pregnancy monitoring by midwives and in zone field conditions:

  * One urban health center (Centralized)
  * One rural health center (Decentralized)
* Assess women's quality of life during pregnancy and obtain satisfaction with echOpen O1 probe.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy ≥ 37 weeks of amenorrhea
* Women aged ≥ 18 years old
* Delivery scheduled to take place in the recruitment center
* Have given her written informed consent to participate

Exclusion Criteria:

* Known fetal morphological abnormality
* Emergency context during the participant's management
* Obstetrical work in progress
* Women anticipating displacement or no delivery at the clinical site

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
The intra-operator agreement | Day 0
  The intra-operator agreement will be measured on the result of the 4 ultrasound targets chosen. The 4 ultrasound targets for each pregnancy are:
  The fetal position; Number of fetuses; Fetal vitality (presence of fetal heartbeat) Placental implantation To define an intra-operator concordance, the images for the 4 ultrasound targets (collected by the same operator) must be identical for both devices (echOpen probe and Ultrasound device routinely used in pregnant women)

SECONDARY OUTCOMES:
The inter-operator agreement | Day 0
  The inter-operator concordance will be measured on the result of the 4 ultrasound targets chosen. The 4 ultrasound targets for each pregnancy are:
  The fetal position; Number of fetuses; Fetal vitality (presence of fetal heartbeat) Placental implantation To define an inter-operator concordance, the images on the 4 ultrasound targets (collected by two different operators) must be identical for the same device (echOpen probe).
  All ultrasound images will go to the radiologist for review and validation. This review will be done blindly of the result provided by the operators.

CONTACTS AND LOCATIONS:
Overall Officials: Fatoumata D. Sarr, M.D., MPH, Principal Investigator — Institut Pasteur de Dakar
Locations (2):
- Senegal (2):
  - Poste de Santé de Karang, Karang, Fatick
  - Centre de Santé de Sokone, Sokone, Fatick

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill CJ, Rowe SI, Lovrien EW. Probable genetic linkage between human serum amylase (Amy 2 ) and Duffy blood group. Nature. 1972 Jan 21;235(5334):162-3. doi: 10.1038/235162a0. No abstract available. PMID 4551225
- [Background] Rundcrantz H. Posture and Eustachian tube function. Acta Otolaryngol. 1969 Oct;68(4):279-92. doi: 10.3109/00016486909121567. No abstract available. PMID 4906986
- [Background] Edvardsson K, Ntaganira J, Ahman A, Sengoma JP, Small R, Mogren I. Physicians' experiences and views on the role of obstetric ultrasound in rural and urban Rwanda: a qualitative study. Trop Med Int Health. 2016 Jul;21(7):895-906. doi: 10.1111/tmi.12718. Epub 2016 May 18. PMID 27125579
- [Background] Tolins SH, Cooper P. Presacral teratoma. Am J Surg. 1968 May;115(5):734-7. doi: 10.1016/0002-9610(68)90114-1. No abstract available. PMID 5645676
- [Background] Ahman A, Edvardsson K, Lesio Kidanto H, Ngarina M, Small R, Mogren I. 'Without ultrasound you can't reach the best decision' - Midwives' experiences and views of the role of ultrasound in maternity care in Dar Es Salaam, Tanzania. Sex Reprod Healthc. 2018 Mar;15:28-34. doi: 10.1016/j.srhc.2017.11.007. Epub 2017 Nov 22. PMID 29389498
- [Background] Gomes DJ, Kaufman B, Aluisio AR, Kendall S, Thomas V, Bloem C. Assessment of Acute Obstetrical Needs and the Potential Utility of Point-Of-Care Ultrasound in the North East Region of Haiti: A Cross-Sectional Study. Ann Glob Health. 2020 Jul 3;86(1):72. doi: 10.5334/aogh.2597. PMID 32676301
- [Background] Glazebrook R, Manahan D, Chater B, Barker P, Row D, Steele B, Morris G, Cornelius S, McLellan T. Educational needs of rural and remote Australian non-specialist medical practitioners for obstetric ultrasound. Aust J Rural Health. 2004 Apr;12(2):73-80. doi: 10.1111/j.1038-5282.2004.00559.x. PMID 15023225
- [Background] Swanson JO, Kawooya MG, Swanson DL, Hippe DS, Dungu-Matovu P, Nathan R. The diagnostic impact of limited, screening obstetric ultrasound when performed by midwives in rural Uganda. J Perinatol. 2014 Jul;34(7):508-12. doi: 10.1038/jp.2014.54. Epub 2014 Apr 3. PMID 24699218
- [Background] Vinayak S, Brownie S. Collaborative task-sharing to enhance the Point-Of-Care Ultrasound (POCUS) access among expectant women in Kenya: The role of midwife sonographers. J Interprof Care. 2018 Sep;32(5):641-644. doi: 10.1080/13561820.2018.1470499. Epub 2018 May 10. PMID 29746179
- [Background] Pound AW, Walker NI. Involution of the pancreas after ligation of the pancreatic ducts. I: a histological study. Br J Exp Pathol. 1981 Dec;62(6):547-58. PMID 7326214
- [Background] Narula J, Chandrashekhar Y, Braunwald E. Time to Add a Fifth Pillar to Bedside Physical Examination: Inspection, Palpation, Percussion, Auscultation, and Insonation. JAMA Cardiol. 2018 Apr 1;3(4):346-350. doi: 10.1001/jamacardio.2018.0001. PMID 29490335
- [Background] Van den Hof MC. No 359-Effets biologiques et innocuite de l'echographie obstetricale. J Obstet Gynaecol Can. 2018 May;40(5):633-639. doi: 10.1016/j.jogc.2018.04.008. No abstract available. PMID 29731209
- [Background] Slavin V, Gamble J, Creedy DK, Fenwick J, Pallant J. Measuring physical and mental health during pregnancy and postpartum in an Australian childbearing population - validation of the PROMIS Global Short Form. BMC Pregnancy Childbirth. 2019 Oct 22;19(1):370. doi: 10.1186/s12884-019-2546-6. PMID 31640626
- [Background] Vinayak S, Sande J, Nisenbaum H, Nolsoe CP. Training Midwives to Perform Basic Obstetric Point-of-Care Ultrasound in Rural Areas Using a Tablet Platform and Mobile Phone Transmission Technology-A WFUMB COE Project. Ultrasound Med Biol. 2017 Oct;43(10):2125-2132. doi: 10.1016/j.ultrasmedbio.2017.05.024. Epub 2017 Jul 14. PMID 28716434
- [Background] Ballard JL, Khoury JC, Wedig K, Wang L, Eilers-Walsman BL, Lipp R. New Ballard Score, expanded to include extremely premature infants. J Pediatr. 1991 Sep;119(3):417-23. doi: 10.1016/s0022-3476(05)82056-6. PMID 1880657
- [Background] Kang C, Qaqish B, Monaco J, Sheridan SL, Cai J. Kappa statistic for clustered dichotomous responses from physicians and patients. Stat Med. 2013 Sep 20;32(21):3700-19. doi: 10.1002/sim.5796. Epub 2013 Mar 27. PMID 23533082
- See also: WHO recommendations on antenatal care for a positive pregnancy experience — https://www.who.int/publications-detail-redirect/9789241549912